CLINICAL TRIAL: NCT00412646
Title: A Randomized, Placebo-controlled Phase II Trial in HIV-1-infected, NRTI-, PI and NNRTI-experienced Subjects to Evaluate the Safety, Tolerability and Efficacy of Different Doses of TMC125 b.i.d. on Top of an Individually Optimized Antiretroviral Therapy by Means of a 2-stage Dose-escalating Design
Brief Title: TMC125-C203: Phase II Randomized (Patients Are Assigned Different Treatments Based on Chance), Placebo Controlled Dose Escalating Trial of TMC125 in HIV-1 Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006754
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Anti-Retroviral Agents; HIV-1
Keywords: HIV; AIDS; Dose finding study; TMC125-C203; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — etravirine

INTERVENTIONS:
Drug: TMC125

SUMMARY:
The purpose of this randomized (patients are assigned different treatments based on chance), placebo-controlled, dose-escalating trial is to evaluate the safety, tolerability and efficacy of different doses of TMC125 twice daily ( b.i.d.) when added to an individually optimized antiretroviral therapy (ART) for 48 weeks. Dose-escalation will be performed in two stages. In the first stage approximately one hundred and eighty HIV-1 positive, three-class ART experienced patients will be randomized to placebo, 400 or 800 mg of TMC125 b.i.d. In the second stage, approximately seventy patients will be randomized to placebo, 800 or 1200 mg TMC125 b.i.d. Stage 2 will be opened for enrollment after review of the available safety and efficacy data for a specified number of patients and concurrence by the Data Safety and Monitoring Board (DSMB). After all patients are treated for a period of 12 weeks, unblinding for the sponsor will occur. The trial will continue in a single-blind fashion (sponsor unblinded, but investigator and patient blinded) for up to 48 weeks. Upon completion of the initial 48 weeks of treatment, patients deriving clinical benefit, in the opinion of the investigator, will have the option to prolong the same treatment, in a single-blind setting up to a maximum of 144 weeks.

DETAILED DESCRIPTION:
Study TMC125-C203 is a phase II, randomized, placebo-controlled, dose-escalating trial that will be conducted in 2 stages. In total approximately two-hundred and fifty HIV-1 positive patients will be included in 2 stages. Patients must be 3-class antiretroviral therapy (ART) experienced (i.e. have previously received at least one protease inhibitor (PI), one nucleoside reverse transcriptase inhibitor (NRTI) and one non-nucleoside reverse transcriptase inhibitor (NNRTI), each for at least 3 months) and must have a VirtualPhenotype™ showing sensitivity to at least 2 antiretroviral drugs used in the optimized underlying ART. Stage 1: approximately 180 patients. 60 patients will receive placebo, 60 patients TMC125 400 mg b.i.d. and 60 patients TMC125 800 mg b.i.d. Stage 2: approximately 70 patients. 10 patients will receive placebo, 20 patients TMC125 800 mg b.i.d. and 40 patients TMC125 1200 mg b.i.d. Screening for study TMC125-C203 will be performed up to six weeks prior to baseline. If a patient fulfills the eligibility criteria he/she will be instructed either not to change his/her current ART until the baseline visit or to continue his/her treatment interruption until baseline. At the baseline visit patients will begin dosing with TMC125 and their optimized ART (composed at the discretion of the investigator), including at least two sensitive antiretroviral drugs as indicated by the VirtualPhenotypeTM. The new optimized underlying ART started at baseline should not be changed until the end of the trial, except for tolerability reasons. Adverse events that begin after the start of study therapy and within 4 weeks after the last dose of study medication will be collected. All adverse events still ongoing at the end of the treatment with TMC125 will be followed until satisfactory resolution or stabilization. Upon completion of the initial 48-week treatment period, patients deriving clinical benefit, in the opinion of the investigator, will have the option to prolong their treatment, with a first optional 48-weeks extension period, followed by a second optional 48-weeks period (maximum treatment duration is 144 weeks). They will continue with the dose of study medication they were assigned to at randomization, in a blinded setting, in addition to their optimized ART initiated during the original treatment period of this study. Four weeks after 120 patients have started treatment in stage 1, all available data will be reviewed by a Data Safety and Monitoring Board (DSMB). Stage 2 will only be opened after concurrence by the DSMB. The primary analysis will be performed once all patients in the two stages have been treated for 24 weeks or have dropped out earlier. The final analysis will be performed when all patients have completed the trial (up to a maximum of 144 weeks), including the follow-up visits, or dropped out earlier. A pharmacokinetic sub-study will be performed within the framework of this trial. The patients enrolled in this sub-study will have additional pharmacokinetic samples taken on top of the assessments described in this protocol to be able to generate a full pharmacokinetic profile of TMC125 and concomitantly administered PIs.The sponsor has the intention to have an open-label follow-up study available for patients who participated in this trial.

Doses of placebo, 400, 800 and 1200 mg TMC125, as twice daily regimens, have been selected for the present trial. The investigational medication will be taken orally every 12 hours and within 15 minutes after breakfast and dinner for 48 weeks (with optional extension period(s) up to a maximum of 144 weeks). All other used underlying antiretroviral drugs will be taken as prescribed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Plasma viral load at screening visit is above 1,000 HIV-1 RNA copies/ml
* Prior use of NRTI, NNRTI and PI, each for at least 3 months
* Currently receiving a stable (for 8 weeks) ART consisting of at least 3 antiretroviral drugs or currently on a treatment interruption for at least 8 weeks
* Further treatment options as defined by sensitivity to at least 2 antiretroviral drugs based on VirtualPhenotype™

Exclusion Criteria:

* Active AIDS defining illnesses
* Patients with a history of severe allergy, hypersensitivity or dermatological manifestation that led to discontinuation while receiving any NNRTI or abacavir
* Pregnant or breast-feeding female
* Female of childbearing potential without the use of effective birth control methods
* Any toxicity above grade 2, except for lipids and glucose, according to the ACTG grading severity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2002-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of different doses of TMC125 b.i.d. (taken twice daily) when added to an individually optimized antiretroviral regimen for 48 weeks.

SECONDARY OUTCOMES:
To evaluate the change in viral load; the proportion of patients with a certain plasma HIV-1 RNA level; the protocol defined virologic endpoints; the degree and duration of immunologic change and the number of patients attaining a virologic response

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Result] Montaner J, Yeni P, Clumeck NN, Fatkenheuer G, Gatell J, Hay P, Seminari E, Peeters MP, Scholler-Gyure M, Simonts M, Woodfall B; TMC125-C203 Study Group. Safety, tolerability, and preliminary efficacy of 48 weeks of etravirine therapy in a phase IIb dose-ranging study involving treatment-experienced patients with HIV-1 infection. Clin Infect Dis. 2008 Oct 1;47(7):969-78. doi: 10.1086/591705. PMID 18764771